CLINICAL TRIAL: NCT04226781
Title: Comparison Between Fluorescenceimaging With Indocyaningreen (ICG) and Hyperspectralimagig (HSI) for Tissue Perfusion in Gastrointestinal Resections
Brief Title: ICG vs. HSI in Gastrointestinal Resections
Acronym: ICGvHSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Boris Jansen-Winkeln, Principal Investigator, Deputy Head of Department, Priv.-Doz. Dr. med. habil., University of Leipzig
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202001
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Anastomosis; Perfusion
Keywords: tissue perfusion; hyperspectral imaging; fluorescence imaging; idocyaningreen (ICG)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG (Active Comparator): Fluorescence imaging for blood Perfusion of the gastrointestinal tissue
  Interventions: Diagnostic Test: Indocyaningreen-Fluorescence imaging
- HSI (Experimental): Hyperspectralimaging for blood Perfusion of the gastrointestinal tissue
  Interventions: Diagnostic Test: Hyperspectral-Imaging

INTERVENTIONS:
Diagnostic Test: Hyperspectral-Imaging — Photos were taken with the hyperspectral camera of the gastrointestinal anastomosis.
  Arms: HSI
Diagnostic Test: Indocyaningreen-Fluorescence imaging — Photos were taken with the Fluorescence camera after injection of the indocyaningreen-dye of the gastrointestinal anastomosis
  Arms: ICG

SUMMARY:
In this study, gastrointestinal anastomoses are examined with a hyperspectral camera and after this the investigators use the Standard Routine ICG-Imaging. At the end, both methods will be compared..

DETAILED DESCRIPTION:
All gastrointestinal anastomoses were examined in all patients with written informed consent.

As Standard in our clinical Routine the tissue perfusion is measured with fluorescence Imaging and Indocyaningreen (ICG). In this study the investigators use the Hyperspectral-Camera (HSI-Camera) as new method. The measurements were performed like described before, using the TIVITA Tissue system (Diaspective Vision GmbH, Am Salzhaff, Germany). This HSI-camera provides hyperspectral images with a high spectral resolution (5 nm) in the visible and near infrared range (500-1000 nm). A RGB image and 4 false color images that represent physiologic parameters are intraoperatively provided by an analysis software. This work is focused on tissue oxygenation (StO2), which represents the relative blood oxygenation in the microcirculation of superficial tissue layers (approximately 1 mm) and the near-infrared (NIR) Perfusion Index, representing tissue layers in 4-6 mm penetration depth.

As Standard method ICG-Fluorescence Imaging is used. After the procedure the Perfusion data of both Systems is compared.

ELIGIBILITY:
Inclusion Criteria:

* all gastrointestinal anastomoses

Exclusion Criteria:

* inability to consent
* allergy against indocyaningreen dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Tissue oxygenation (StO2) in % | After the intraoperative Photo is taken, within 5 minutes
  Directly after the photo has been taken, the distribution of the spectra and their intensity is evaluated with the help of computer assisted analysis software. The software calculates the tissue oxygen saturation value (StO2) in percent. These values are measured at a standardized distance from the anastomosis region.
Anastomotic Perfusion in arbitrary units | After the intraoperative Photo is taken, within 5 minutes
  Directly after the photo has been taken, the distribution of the spectra and their intensity is evaluated with the help of computer assisted analysis software. The software calculates the tissue perfusion in arbitrary units. (Method is described in attached literature) These values are measured at a standardized distance from the anastomosis region.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Jansen-Winkeln, MD, PD, Principal Investigator — University of Leipzig
Locations (1):
- Universitätsklinikum Leipzig - AöR, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
no sharing

REFERENCES:
- [Background] Jansen-Winkeln B, Holfert N, Kohler H, Moulla Y, Takoh JP, Rabe SM, Mehdorn M, Barberio M, Chalopin C, Neumuth T, Gockel I. Determination of the transection margin during colorectal resection with hyperspectral imaging (HSI). Int J Colorectal Dis. 2019 Apr;34(4):731-739. doi: 10.1007/s00384-019-03250-0. Epub 2019 Feb 2. PMID 30712079
- [Background] Jansen-Winkeln B, Maktabi M, Takoh JP, Rabe SM, Barberio M, Kohler H, Neumuth T, Melzer A, Chalopin C, Gockel I. [Hyperspectral imaging of gastrointestinal anastomoses]. Chirurg. 2018 Sep;89(9):717-725. doi: 10.1007/s00104-018-0633-2. German. PMID 29637244
- [Derived] Jansen-Winkeln B, Germann I, Kohler H, Mehdorn M, Maktabi M, Sucher R, Barberio M, Chalopin C, Diana M, Moulla Y, Gockel I. Comparison of hyperspectral imaging and fluorescence angiography for the determination of the transection margin in colorectal resections-a comparative study. Int J Colorectal Dis. 2021 Feb;36(2):283-291. doi: 10.1007/s00384-020-03755-z. Epub 2020 Sep 23. PMID 32968892